CLINICAL TRIAL: NCT05796791
Title: Ketamine and Motivational Enhancement Therapy for the Treatment of Tobacco Use Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00126022
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Tobacco Use; Smoking Cessation; Nicotine Dependence
MeSH Terms: conditions — Tobacco Use; Smoking Cessation; Tobacco Use Disorder | interventions — Ketamine; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Pilot Study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment of tobacco use disorder with ketamine (Experimental)
  Interventions: Drug: Ketamine Hydrochloride; Behavioral: Motivational enhancement therapy

INTERVENTIONS:
Drug: Ketamine Hydrochloride — IM ketamine given in weekly session for a total of 3 weeks
Behavioral: Motivational enhancement therapy — Brief motivational based therapy

SUMMARY:
The purpose of the study is to examine whether an investigational medication called ketamine is able to improve treatment outcomes for tobacco use disorder when delivered in conjunction with brief motivational enhancement therapy. Participants will receive ketamine assisted motivational enhancement therapy weekly for three weeks and there will be 2 follow up visits. All visits will also consist of questionnaires and saliva samples will be taken. The overall participation will last approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 21 to 65 years old.
2. Able to provide informed consent.
3. Be a daily cigarette smoker with multiple unsuccessful previous quit attempts, and report a continued desire to quit smoking.
4. Agree to abstain from smoking for the ketamine session from 1 hour before ketamine administration
5. Agree to refrain from using any psychoactive drugs, including alcoholic beverages, within 24 hours of ketamine administration. Exceptions include caffeine and nicotine.
6. Subjects taking other psychotropic medications must be maintained on a stable dose for at least four weeks before study initiation.
7. Be healthy as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG) to verify normal QTc intervals.
8. Subjects with normal blood pressure not on antihypertensive medications or medication controlled hypertension as defined baseline visit systolic blood pressure (SBP) <140 mmHg or a diastolic blood pressure (DBP) <90 mmHg.

Exclusion Criteria:

1. Women who are pregnant (positive pregnancy test) or nursing, or are not practicing an effective means of birth control which can include oral, implant, intrauterine device, or patch contraceptive methods as well as barrier contraceptive methods, history of surgery such as hysterectomy or tubal ligation, or abstinence
2. Subjects who meet DSM-5 criteria for current or history of psychotic spectrum disorders or current depression or bipolar disorder based on clinical interview.
3. Subjects meeting DSM-5 criteria for current substance use disorder other than tobacco use disorder.
4. Subjects with hypertension as defined by a baseline visit systolic blood pressure (SBP) >140 mmHg or a diastolic blood pressure (DBP) >90 mmHg.
5. A history of allergic or other adverse reaction to ketamine (or its excipients).
6. Clinically significant physical exam findings or self-reported medical conditions for which a transient increase in blood pressure could be significantly detrimental (e.g. glaucoma, aneurysmal disease, cardiovascular disease, or end-stage renal disease).
7. Cardiovascular conditions: uncontrolled hypertension, angina, a clinically significant ECG abnormality (e.g., atrial fibrillation), TIA in the last 6 months, stroke, peripheral or pulmonary vascular disease
8. Subjects who live greater than 20 miles from the study site and cannot arrange their own transportation will be excluded from the study.
9. Subjects with clinically significant kidney or liver impairment.
10. Have any current neurological illnesses including, but not limited to, seizure disorders, frequent migraines or on prophylaxis, multiple sclerosis, movement disorders, history of significant head trauma, or CNS tumor.
11. Morbidly obese (BMI >40), or severely underweight as determined by medical examination.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment of Tobacco Use Disorder With Ketamine
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Number of subjects enrolled.
Arm/Group | Treatment of Tobacco Use Disorder With Ketamine
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Ketamine Treatment for Tobacco Use Disorder
Description: The primary outcome of this study will be the feasibility of using ketamine-assisted treatment for smoking cessation, which will assess the number of people selected for randomization that complete the full treatment. This will help determine if the treatment of ketamine in tobacco use would be beneficial for further study.
Time Frame: 8 weeks
Population: Number of participants enrolled that completed all three interventional sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of Tobacco Use Disorder With Ketamine
Number analyzed (Participants) | 7
Participants | 7

2. Secondary Outcome: Smoking Cessation
Description: Saliva cotinine levels will be collected prior to each ketamine session and at each follow up to detect smoking over approximately the past 6 days
Time Frame: Baseline, Treatment week 1, 2, 3, and follow up week 4, and 8
Reporting Status: Not Posted

3. Secondary Outcome: Reduction in Cigarettes Smoked Per Day
Description: Evaluate if there is reduction in cigarettes smoked per day via the self-reported time-line follow back
Time Frame: Baseline, Treatment week 1, 2, 3, and follow up week 4, and 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 1 year
Groups:
- Treatment of Tobacco Use Disorder With Ketamine: No adverse event outcome
Arm/Group | Treatment of Tobacco Use Disorder With Ketamine
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT05796791/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT05796791/ICF_000.pdf